CLINICAL TRIAL: NCT07353697
Title: Evaluation of the Effects of Different Therapeutic Play Methods on Pre- and Post-operative Anxiety and Acute Symptoms in School-aged Children Aged 6-12
Brief Title: Evaluation of Therapeutic Play Methods on Preoperative Anxiety and Acute Postoperative Symptoms in School-Age Children
Acronym: TP-MAPAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E-10333602-050.04-253950
Record Dates: First submitted 2025-12-29; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Preoperative Anxiety; Postoperative Complications
Keywords: Pediatric surgery; play therapy; virtual reality; anxiety
MeSH Terms: conditions — Postoperative Complications; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard Maintenance (No Intervention): This arm includes children who did not receive any therapeutic play intervention during the preoperative period and only underwent the standard clinical preparation process.
- Finger Puppet Therapeutic Game (Experimental): This arm includes children who participated in the structured finger puppet therapeutic play activity administered by the researcher during the preoperative period. The intervention involves interaction with age-appropriate puppets and guided play-based distraction techniques.
  Interventions: Other: Finger Puppet Play
- Virtual Reality (VR) Game (Experimental): This arm includes children who participated in an interactive VR game experience using virtual reality goggles during the preoperative period. The intervention is based on visual and auditory stimuli aimed at distracting the child's attention from the surgical process.
  Interventions: Other: Virtual Reality Play
- Smartphone-Based Game (Experimental): This arm includes children who experience distraction and game-focused interaction guided by an age-appropriate smartphone game during the preoperative period.
  Interventions: Other: Smartphone Game Play

INTERVENTIONS:
Other: Finger Puppet Play — Finger Puppet Play - Intervention Description This intervention is a guided therapeutic play activity that involves the child interacting with age-appropriate finger puppets during the preoperative period. The application is conducted by the researcher according to a standard protocol and combines imaginative play with attention-focused play techniques. The intervention aims to regulate the child's emotions, divert their attention away from the surgical process, and create a relaxing play environment through puppet characters.
  Arms: Finger Puppet Therapeutic Game
Other: Virtual Reality Play — Virtual Reality Play - Intervention Description This intervention involves directing the child to an age-appropriate visual-auditory gaming experience through virtual reality goggles. VR content provides interactive environments designed to distract the child's attention away from the surgical process. The application is carried out for a fixed period of time and according to a standardized protocol. The intervention is a technology-based distraction technique that aims to reduce anxiety and tension by providing multi-sensory stimulation.
  Arms: Virtual Reality (VR) Game
Other: Smartphone Game Play — Smartphone Game Play - Intervention Description This intervention is based on the child playing an age-appropriate smartphone game selected by the researcher during the preoperative period. The application uses one-way or interactive game content and is carried out for a standard period of time. The intervention is designed as an easily accessible digital distraction method and aims to divert the child's cognitive focus away from the surgical process.
  Arms: Smartphone-Based Game

SUMMARY:
This study aims to evaluate the effect of different therapeutic play methods (finger puppet play, virtual reality glasses, and smartphone games) applied to children aged 6-12 years during the preoperative period on their anxiety levels and postoperative acute symptoms. The study has a randomized controlled design conducted in a pediatric surgery clinic. The research seeks to answer the following question: "Are different therapeutic play methods effective in reducing anxiety, fear, pain, and other acute symptoms in children during the surgical process?"

DETAILED DESCRIPTION:
Psychological stress experienced by children prior to surgical intervention can increase autonomic nervous system activation, thereby affecting pain perception, nausea development, hemodynamic variability, and the recovery process during the perioperative period. Therapeutic play interventions are non-invasive interventions that support children's coping skills with the surgical process through mechanisms such as distraction, cognitive restructuring, and emotional regulation. In recent years, technology-based approaches such as virtual reality have begun to be used in pediatric surgery as an alternative or complementary component to traditional play methods. However, randomized controlled data comparing the effects of these methods on physiological and psychological responses are still limited.

This study employs an experimental design aimed at examining the capacity of different game-based interventions administered during the preoperative period to regulate children's stress response. The intervention protocols target different mechanisms, including visual-auditory stimulation, cognitive attention guidance, imaginative play, and the use of interactive digital stimuli. Physiological changes are monitored at standardized time points, and early responses of the autonomic response (heart rate, blood pressure, breathing pattern) to game-based distractions are recorded for evaluation. Psychological assessments are structured to measure the child's emotional regulation capacity, anxiety level, and behavioral responses during the surgical process in a multidimensional manner.

Additionally, the study includes an assessment of the perioperative care experience from the family perspective. This assessment aims to understand the potential indirect effects of play interventions on parent-child interaction, parental trust in healthcare, and parental involvement in the care process. The multi-arm design of the study allows for the comparison of different therapeutic play techniques and the determination of which intervention potentially has a stronger effect on specific clinical outcomes.

The data obtained in this context aims to reveal the applicability, clinical effect profiles, and potential areas of application of play-based interventions for non-pharmacological anxiety management in pediatric surgical practice.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 12 years
* Hospitalized at Bilecik Training and Research Hospital, Department of Pediatric Surgery, for an elective surgical procedure
* Able to read and write
* Able to communicate in Turkish
* No visual, hearing, or speech impairments
* No intellectual disability or physical or surgical condition that would interfere with participation
* Voluntary participation with written informed consent obtained from the child and the parent or legal guardian

Exclusion Criteria:

* Children referred to the intensive care unit
* Children requiring repeat surgical intervention
* Children with a hospital stay of two days or longer
* Children with severe psychiatric disorders

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
Changes in State Anxiety Scores in Children During the Preoperative Period | Preoperative baseline (Day 0); immediately after the preoperative therapeutic play intervention (Day 0, before surgery); 2 hours after surgery (Day 0); approximately 30 minutes before discharge (Day 1)
  Anxiety level is assessed using the State Anxiety Inventory for Children, which consists of 20 items with total scores ranging from 20 to 60. Higher scores indicate higher levels of anxiety, whereas lower scores indicate lower levels of anxiety. Anxiety assessments are conducted at four time points: preoperative baseline (Day 0); immediately after the preoperative therapeutic play intervention (Day 0, before surgery); 2 hours after surgery (Day 0); and approximately 30 minutes before discharge (Day 1).

CONTACTS AND LOCATIONS:
Overall Officials: Dilek AYGİN, PROF. DR, Principal Investigator — Sakarya University
Locations (1):
- Bilecik Training and Research Hospital, Bilecik, Bilecik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) collected as part of the study will not be shared due to the inclusion of sensitive personal health information of child participants and the risk of re-identification. Access to IPD is restricted in accordance with data confidentiality and ethical requirements.